CLINICAL TRIAL: NCT05825599
Title: An Interventional, Non-comparative, Single-center Post Marketing Clinical Follow-up (PMCF) Study to Evaluate Performance and Safety of "Hydroxypropyl Methylcellulose (HPMC)-Based Eyedrops" Used to Relieve Dry Eye Symptoms
Brief Title: PMCF Study to Evaluate Performance and Safety of "HPMC-based Eyedrops" Used to Relieve Dry Eye Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C.O.C. Farmaceutici S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COC-R3-HPMC
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Dry Eye; Dry Eye Disease; Kerato Conjunctivitis Sicca
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eyedrops treatment arm (Experimental)
  Interventions: Device: Hydroxypropyl methylcellulose eye drops

INTERVENTIONS:
Device: Hydroxypropyl methylcellulose eye drops — Hydroxypropyl methylcellulose (HPMC)-based eyedrops

SUMMARY:
Dry eye disease (DED), also called keratoconjunctivitis sicca, is a common ocular condition characterized by a loss of homeostasis of the tear film and inflammation of the ocular surface.

Over the counter (OTC) artificial tears are typically the first line of dry eye treatment; they are meant to supplement the tears that cover the eye's surface. OTC products mimic the different layers of the tear film in order to maintain ocular hydration.

Hydroxypropyl methylcellulose (HPMC or hypromellose) is a synthetic modification of the natural polymer, cellulose. It has been widely used in in ophthalmologic formulations such as eye drops and gels due to its solubility in water, biocompatibility, transparency and rheological properties. Eye drops containing HPMC are conventionally used to treat tear film disturbances including dry eye symptoms.

For these reasons, an interventional, non-comparative, single-center Post Marketing Clinical Follow-up (PMCF) study was planned to evaluate the performance and safety of "Hydroxypropyl methylcellulose (HPMC)-based eyedrops" used as intended to relieve dry eye symptoms.

The objectives of the PMCF study are confirmation of the performance, collection of additional safety data regarding expected adverse events and detection of potential unexpected adverse events associated with use of "HPMC-based eyedrops" according to the Instructions for Use (IFU).

"HPMC-based eyedrops" medical devices are ophthalmic solutions containing hydroxypropyl methylcellulose (HPMC) as key ingredient, a polymer able to relief eye discomfort thanks to its moisturizing, lubricating and muco-mimetic properties. HPMC can stabilize the tear film on the ocular surface by creating a protective, transparent and viscoelastic shield.

Each subject, after signing the Informed Consent Form (ICF), will enter the screening and baseline phase (the 2 visits will coincide) during which baseline procedures will be completed.

At baseline visit (V0), only one of the below reported "HPMC-based eyedrops" products will be administered to the enrolled subject.

The patient will perform 2 on-site visits: V0 and V2/EOS. To monitor the safety, 1 phone contact is planned (V1) to check for potential adverse events and concomitant medications intake.

ELIGIBILITY:
Inclusion Criteria:

* Patient Informed consent form (ICF) signed;
* Male and Female Aged ≥ 18 years at the time of the signature of the ICF;
* Patients with ocular symptoms such as burning, itching, and foreign body sensation due to environmental factors, contact lenses wearing, and/or moderate-severe dry eye symptoms;
* Willing not to use other eye drops during the entire treatment period.

Exclusion Criteria:

* Other - different - eyes clinical conditions (e.g. glaucoma);
* Suspected alcohol or drug abuse.
* Known hypersensitivity or allergy to Investigational Product (IP) components;
* Other clinically significant and uncontrolled pathologies that may interfere with study results (e.g. rheumatic diseases, diabetes);
* Participation in another investigational study;
* Inability to follow all study procedures, including attending all site visits, tests and examinations;
* Mental incapacity that precludes adequate understanding or cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Change in Schirmer Test I: to evaluate the performance of the "HPMC-based eyedrops" used to relieve dry eye symptoms by moisturizing and lubricating the ocular surface, through Schirmer I test | From baseline (V0 = Day 0) to 1 month (EOS/V2 = Day 30)

SECONDARY OUTCOMES:
Change in Ocular Surface Disease Index (OSDI): to evaluate the performance of the "HPMC-based eyedrops" used to provide soothing and refreshing relief in subjects with eye discomfort sensation, through OSDI | From baseline (V0 = Day 0) to 1 month (EOS/V2 = Day 30)
Change in Tear Break-up Time (TBUT): to evaluate the protecting eye-surface performance of the "HPMC-based eyedrops" by stabilizing the tear film in subjects with moderate dry eye or severe dry eye, through the TBUT test | From baseline (V0 = Day 0) to 1 month (EOS/V2 = Day 30)
To evaluate the safety and tolerability of the "HPMC-based eyedrops" through Visual Analogue Scale (VAS) - evaluation of symptoms related to dry eye disease (burning, fatigue, discomfort, redness) | End of study visit (EOS/V2 = Day 30)
  Visual Analogue Scale:
  Minimum value = 0; Maximum value = 10; Higher scores mean a better outcome.
To evaluate the patient satisfaction of the "HPMC-based eyedrops" through a 5-points Likert Scale | End of study visit (EOS/V2 = Day 30)

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Policlinico Mater Domini - Università Magna Grecia di Catanzaro, Catanzaro, CZ, Italy